CLINICAL TRIAL: NCT01171066
Title: Assessment of the Performance of the Tasman CPAP System in Treating Obstructive Sleep Apnea
Brief Title: Performance of the Tasman Continuous Positive Airway Pressure (CPAP) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA14010
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tasman CPAP (Experimental)
  Interventions: Device: Tasman CPAP system

INTERVENTIONS:
Device: Tasman CPAP system — Participants will trial the Tasman CPAP system for a duration of 1 week in place of their current CPAP system.
  Other Names: ResMed Tasman

SUMMARY:
Assessment of the performance of the Tasman CPAP system in treating obstructive sleep apnea. The purpose of this study is to (1) evaluate the performance of this system in the efficacy of the treatment in comparison to S8 Escape, and (2) to evaluate the performance of the Tasman device via subjective assessment of comfort and ease of breathing compared to the participant's current CPAP device.

DETAILED DESCRIPTION:
Obstructive Sleep Apnoea (OSA) is a condition characterised by partial or complete collapse of the upper airway during sleep. The treatment of choice for OSA is Continuous Positive Airway Pressure (CPAP). CPAP acts as a positive airway splint, delivering a fixed positive airway pressure to the upper airway via a tube and mask. The mask is attached to the participant's nose via head straps. The type of mask used is dependent upon participant choice and comfort and the mask that provides the best fit.

Some participants stop using CPAP therapy finding it difficult to tolerate due to leak issues or discomfort from their nasal mask. Another frequent concern is mask dislodgment while sleeping causing leaks and consequently waking the patient up.

The purpose of this study is to evaluate the performance of the Tasman CPAP system via objective and subjective assessment of comfort and ease of breathing compared to the participant's current CPAP device.

Aim

* To determine if the efficacy of the treatment is clinically equivalent to or better than the predicate device (S8 Escape)
* To evaluate the performance of the Tasman CPAP system in terms of comfort of breathing and general ease of use

ELIGIBILITY:
Inclusion Criteria

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients being treated for OSA for >6 months
* Patients using a ResMed nasal mask system
* Patients who can trial the trial mask for 7 nights

Exclusion Criteria

* Patients not willing to give written informed consent
* Patients who can not read and comprehend English
* Patients being treated for OSA for <6 months
* Patients using an inappropriate mask system
* Patients using Bilevel flow generators
* Patients who are not using CPAP between 7 and 13 cmH2O
* Patients who are pregnant
* Patients who cannot trial the trial mask for 7 nights
* Patients with a hearing impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To determine if the efficacy of the treatment is clinically equivalent to or better than the predicate device (S8 Escape) | 1 week

SECONDARY OUTCOMES:
To assess the usability of the Tasman CPAP system | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, Principal Investigator — ResMed
Locations (1):
- ResMed Ltd, Sydney, New South Wales, Australia